CLINICAL TRIAL: NCT06100458
Title: Use of Skin and Leakage Protocol and Its Impact on Continence Care at Nursing Homes in the UK.
Brief Title: Use of Continence Care Protocol in UK Nursing Homes.
Status: Completed | Type: Observational
Sponsor: Essity Hygiene and Health AB (Industry)
Collaborators: Lincolnshire Community Health Services NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LASTER
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Urinary Incontinence Due to Cognitive Impairment; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Protocol arm: The skin and leakage protocol was used over a 5 day baseline period. The follow up was done 25 days later by another 5 day period of protocol use to observe any changes in continence care.
  Interventions: Other: Skin and leakage protocol

INTERVENTIONS:
Other: Skin and leakage protocol — The skin and leakage protocol have been developed by the sponsor with the aim to offer a tool that can aid care providers in identifying problems in continence care and follow up the effect of any care interventions to remedy these problems. The protocol is a digital diary tool that tracks both the instances of urine leaking out of an absorbing incontinence product onto clothes and bedsheets, and any apparent skin changes in the area covered by the product. The protocol is in clinical use at the care homes were the subjects are residing.

SUMMARY:
This is a retrospective cohort study. In the investigation the clinical use of the Skin and leakage protocol (SLEP) is to be investigated. The SLEP is a generic digital diary form filled out to give information about the current status of continence care among care home residents. The SLEP tracks the number of leakage occurrences and daily skin health over a period of time with the purpose of assisting care staff in making decisions regarding continence care. The SLEP has been introduced at several United kingdom National Health Service care homes and with this investigation the investigators want to retrospectively analyse the data to determine the clinical usefulness of the form.

The primary objective of the study is to describe any changes in product leakage rate at the baseline and follow up time period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with urinary incontinence managed with an absorbing incontinence product.
* The skin and leakage protocol have been used in the care of the subject and there is data from at least two measurements.
* Subject is cared for in a Residential care home using the skin and leakage protocol.
* Subject is over 18 years of age.

Exclusion Criteria:

* Subject is not using an absorbing incontinence product to manage incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be evaluated will be subjects of the selected Care homes who meet all the required Inclusion and Exclusion criteria and who's data is available on the appropriate databases. Subjects will be considered eligible to participate in the study if:
  All eligible subjects, that data is available for, cared for at the selected care homes and subjected to the protocol are to be assessed. Typically, all residents that use containment products are assessed at the care home.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Change in leakage rate | 28 days
  Change in absorbing product leakage rate between baseline and follow up period

SECONDARY OUTCOMES:
Subject care profile | 28 days
  The care needs profiles of the subjects using the skin and leakage protocol. According to specific criteria for degree of confusion and mobility subjects can be assigned one of 6 different profiles. The profiles are arranged on a scale from 1-6 were 1 is lowest level of care need and 6 is the highest.
Change in skin health score | 28 days
  Change in skin health assessment score between the baseline and follow up period. The skin assessment is conducted on a scale from 1-5 were 1 represents no presence of skin irritation and 5 represents severe skin problems.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Jeffrey, Principal Investigator — Lincolnshire Community Health Services National Health Services Trust
Locations (1):
- Lincolnshire Community Health Services NHS Trust, Lincoln, United Kingdom